CLINICAL TRIAL: NCT04031820
Title: Effectiveness of Dual-mobility Cups for Preventing Dislocation After Primary Total Hip Arthroplasty by a Posterolateral Approach and Their Cost-effectiveness Compared to Unipolar Cups in Elderly Patients.
Brief Title: Dual-mobility Cups Compared to Unipolar Cups on Dislocation and Cost-effectiveness After Primary Total Hip Arthroplasty.
Acronym: REDEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JointResearch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL64819.100.18
Record Dates: First submitted 2019-01-10; First posted 2019-07-24 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Total Hip Arthroplasty; Osteoarthritis, Hip
Keywords: Primary total hip arthroplasty; Dual Mobility cup
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- unipolar cup (Active Comparator): 550 patients will receive a total hip arthroplasty with a unipolar cup.
  Interventions: Procedure: Unipolar cup
- Dual Mobility cup (Active Comparator): 550 patients will receive a total hip arthroplasty with a dual mobility cup.
  Interventions: Procedure: Dual mobility cup

INTERVENTIONS:
Procedure: Unipolar cup — Cemented unipolar acetabulum cup for primary THA
  Arms: unipolar cup
Procedure: Dual mobility cup — Cemented dual mobility acetabulum cup for primary THA
  Arms: Dual Mobility cup

SUMMARY:
Objective: The primary objective is to investigate whether there is a difference in the number of hip dislocations following primary total hip arthroplasty (THA), using the posterolateral approach, with a DM cup compared to a unipolar cup in elderly patients 1 year after surgery.

Study design: Prospective multi-center nation wide, single blinded RCT nested in the LROI.

Study population: Patients ≥ 70 years old, undergoing an elective primary cemented THA.

DETAILED DESCRIPTION:
Rationale: Dislocation is the leading reason for early revision surgery. To address the problem of dislocation, the dual-mobility (DM) cup was developed in France in the 1970's. This cup should provide more stability and biomechanically reduce the risk of dislocation. In the Netherlands, most DM cups are placed in specific patients, e.g. with cognitive impairment and for revisions due to recurrent dislocations. Despite the increased and, in some countries, broad use of DM cups, high quality evidence of their (cost)effectiveness is lacking. This study aims to perform a trial to fill this gap in knowledge. Much of the information needed to judge the effectiveness of DM cups is already incorporated in the Dutch Arthroplasty Register (LROI). This register lends itself perfectly for a nested RCT towards this aim.

Objective: The primary objective is to investigate whether there is a difference in the number of hip dislocations following primary total hip arthroplasty (THA), using the posterolateral approach, with a DM cup compared to a unipolar cup in elderly patients 1 year after surgery. The secondary objectives are: to investigate whether there is a difference in the number of revisions; to investigate what the cost-effectiveness and cost-utility is of a DM cup compared to a unipolar cup at 1 year follow-up; to investigate whether there is a difference in the number of hip dislocations and revisions between a DM cup and a unipolar cup 2 years after surgery; to investigate whether there is a difference in patient reported outcomes between a DM cup compared to a unipolar cup 1 and 2 years after surgery; to compare the number of hip dislocations, revisions and PROM data between patients in the randomized DM group and patients in an observational cohort DM group. Finally, long-term survival of DM and unipolar cups will be evaluated based on revision and mortality data registered in the LROI.

Study design: Prospective multi-center nation wide, single blinded RCT nested in the LROI.

Study population: Patients ≥ 70 years old, undergoing an elective primary cemented THA.

Intervention (if applicable): The intervention group receives a THA with a dual mobility cup, the control group receives a THA with a unipolar cup.

Main study parameters/endpoints: Primary: The number of dislocations. Secondary: costs, patient reported outcomes and implant survival.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In addition to the benefits from regular care, the primary hip arthroplasty procedure, patients might benefit from randomization to receiving a DM cup. DM cups are designed to reduce the risk of hip dislocation, compared to a unipolar cup. Patients may undergo more thorough follow-up than non-study patients and may benefit from this increased surveillance compared with regular care. The only burden associated with study participation is the time needed to complete the cost questionnaires (all other outcomes are part of standard care).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for elective primary THA with a cemented cup, with a 32mm or 36 mm liner, for any indication.
* THA using posterolateral surgical approach.
* Patients ≥ 70 years old
* Adequate comprehension of written and spoken Dutch

Exclusion Criteria

* Patients unable to complete PROMs
* Patients with dementia, epilepsy*, spasticity*, mental retardation or alcoholism. (If dementia or mental retardation is not already mentioned in the medical chart, this can be determined by doctors opinion.)
* Patients not eligible for either a unipolar or a DM cup

  * These patients will be asked to participate in the non-randomized dual mobility observational cohort.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of dislocations | 1 year postoperative
  The total number of dislocations, regardless of type of treatment (i.e. closed repositioning or revision).

SECONDARY OUTCOMES:
Number of revision surgeries | 1 year postoperative
  Revision surgery of any component for any reason
cost-effectiveness questionnaire | 1 year postoperative
  An economic evaluation will be performed from the societal perspective, for dislocation and Quality Adjusted Life Years (QALYs). Prevailing guidelines of Zorginstituut Nederland will be observed. All costs and consequences relevant to THA, hip dislocation and hip revision will be taken into account. To compare costs between groups, confidence intervals around the mean differences in costs at one year after THA will estimated using the bias-corrected and accelerated bootstrap method.
Number of dislocations | 2 years postoperative
  Total number of dislocations
Patient Reported Outcomes on physical functioning | 1 and 2 years postoperative
  Difference in patient reported outcomes on physical functioning following primary THA with a DM cup compared to a unipolar cup, measured with the Hip disability and Osteoarthritis Outcome Score Physical Short form (HOOS-PS). Interval level scores from 0 (no difficulty) to 100 (extreme difficulty).
Patient Reported Outcomes on pain | 1 and 2 years postoperative
  Difference in patient reported outcomes on pain, following primary THA with a DM cup compared to a unipolar cup, measured with the Numeric Ratin Scale (NRS) for pain in rest and during weight bearing. 0 means no pain, 10 means the most extreme pain.
Patient Reported Outcomes on quality of life | 1 and 2 years postoperative
  Difference in patient reported outcomes quality of life, following primary THA with a DM cup compared to a unipolar cup, measured with the EuroQol 5 Dimensions (EQ-5D). A higher score means a worse quality of life, a lower score means a better quality of life. For the visual analogue scale (part of the EQ-5D), the lowest means the worst an the highest score means the best health score.
Implant survival | 5 - 10 years postoperative
  Long-term implant survival based on LROI revision and mortality data.

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Poolman, MD, PhD, Principal Investigator — OLVG, Amsterdam, the Netherlands
Locations (1):
- OLVG, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Beers LWAH, Van Der Wal BCH, Van Loon TG, Moojen DJF, Van Wier MF, Klaassen AD, Willigenburg NW, Poolman RW; Collaborator group. Study protocol: Effectiveness of dual-mobility cups compared with uni-polar cups for preventing dislocation after primary total hip arthroplasty in elderly patients - design of a randomized controlled trial nested in the Dutch Arthroplasty Registry. Acta Orthop. 2020 Oct;91(5):514-519. doi: 10.1080/17453674.2020.1798658. Epub 2020 Aug 4. PMID 32746668